CLINICAL TRIAL: NCT05219396
Title: The Comparison of Proprioception and Gait Function Among Different Rotational Designs in Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMUH110-REC2-235
Record Dates: First submitted 2022-01-19; First posted 2022-02-02 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Arthroplasty, Replacement, Knee; Proprioception; Gait; Balance
Keywords: knee arthroplasty; rotational design; proprioception; balance function; gait performance
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- mobile bearing (MB)
  Interventions: Device: Knee arthroplasty
- medial congruent (MC)
  Interventions: Device: Knee arthroplasty
- posterior stabilized (PS)
  Interventions: Device: Knee arthroplasty

INTERVENTIONS:
Device: Knee arthroplasty — Your knee should be replaced with mobile bearing (MB), medial congruent (MC) and posterior stabilized (PS) design protheses.

SUMMARY:
The symptoms of knee osteoarthritis include knee joint pain, impaired proprioception, and etc. Knee arthroplasty is commonly recommended for the patient with severe knee osteoarthritis to relieve pain and regain function. But the effects of arthroplasty on the proprioception and gait performance, which were related to the risk of falling, were not fully understood. Recently, the concept of enhancing the rotational movement has been introduced into the design of the knee joint prosthesis for mimicking the kinematic performance of the healthy knee. However, study on the functional performance after using these rotational designed arthroplasties was still scarce. So, the purpose of this study aims to evaluate the differences in the proprioception, balance function and gait performance among different designs of the knee arthroplasties with mobile bearing (MB), medial congruent (MC) and posterior stabilized (PS) design. This study is divided into the retrospective and prospective parts.

Investigators will enroll the patients who already replaced their knee joint by one of the above knee arthroplasties for the retrospective part; other patients who plans to receive one of the above knee arthroplasties, twenty participants for each design and each part. The assessment of proprioception, balance function and gait performance will be performed before the knee arthroplasty, and followed at the post-surgery time points of six weeks and three months. The one-way ANOVA will be used to compare the group differences in the retrospective part, and the two-way mixed model ANOVA for the prospective part.

Ultimately, the results of this study could help to have better knowledge of the treatment effects from the different designed knee arthroplasties.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as knee joint osteoarthritis and will receive knee joint arthroplasty.

Exclusion Criteria:

* Already receiving a knee joint arthroplasty surgery
* Can not walk independently for 20 m
* Can not stand for 5 min
* With neurological degenerative disease
* Lower limb received any surgery within recent 2 years

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out patient department
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
Knee joint proprioception | Pre-operation
  Degrees
Knee joint proprioception | Post-operation 6 weeks
  Degrees
Knee joint proprioception | Post-operation 3 months
  Degrees
Postural stability index | Pre-operation
  Degrees
Postural stability index | Post-operation 6 weeks
  Degrees
Postural stability index | Post-operation 3 months
  Degrees
Angle of foot during walking | Pre-operation
  Degrees
Angle of foot during walking | Post-operation 6 weeks
  Degrees
Angle of foot during walking | Post-operation 3 months
  Degrees
Western Ontario and McMaster Universities Osteoarthritis Index, WOMAC | Pre-operation
  Scoring from 0 to 100, and higher scores mean a better outcome.
Western Ontario and McMaster Universities Osteoarthritis Index, WOMAC | Post-operation 6 weeks
  Scoring from 0 to 100, and higher scores mean a better outcome.
Western Ontario and McMaster Universities Osteoarthritis Index, WOMAC | Post-operation 3 months
  Scoring from 0 to 100, and higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No